CLINICAL TRIAL: NCT01048294
Title: Gerandomiseerde en Gecontroleerde Studie Naar de Effecten Van Lichttoediening Met Een Hogere Kleurtemperatuur in Vergelijking Met de Standaard Lichttherapie in de Behandeling Van Winterdepressie
Brief Title: Blue Enriched Versus Standard Light Treatment for Seasonal Affective Disorder(SAD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Ybe Meesters, PhD, University Medical Center Groningen
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: METc2005/160
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2005-10

CONDITIONS: Seasonal Affective Disorder
Keywords: Seasonal affective disorder; phototherapy; circadian rhythms; blue enriched light; melanopsin; Primary disease: Seasonal Affective Disorder, winter type
MeSH Terms: conditions — Seasonal Affective Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Light Treatment (Active Comparator): 30 min of Standard bright light treatment (color 5000K)
  Interventions: Device: Original Energy Light,
- Blue enriched Light treatment 20 min (Experimental): 20 minutes of Blue enriched light treatment (color 17000K)
  Interventions: Device: Original Energy Light prototype
- Blue enriched light treatment 30 min (Experimental): 30 minutes of Blue enriched light treatment (color 17000K)
  Interventions: Device: Original Energy Light prototype

INTERVENTIONS:
Device: Original Energy Light, — 9000 lux, 30 minutes in the morning
  Other Names: Philips energy light HF 3308; 2 lamps PLL36W color 5000K
  Arms: Standard Light Treatment
Device: Original Energy Light prototype — 9000 lux 20 minutes in the morning
  Other Names: Philips energy light HF 3308; 2 lamps PLL36W color 17000K
  Arms: Blue enriched Light treatment 20 min
Device: Original Energy Light prototype — 9000 lux 30 minutes in the morning
  Other Names: Philips energy light HF 3308; 2 lamps PLL36W color 17000K
  Arms: Blue enriched light treatment 30 min

SUMMARY:
One of the most frequently investigated hypothesis of the pathophysiology underlying Seasonal Affective Disorder(SAD) or so called winterdepression is a disturbance of circadian rhythms. Since the circadian system is especially sensitive for the blue portion of the light spectrum, a new light therapy device with more blue light (blue enriched polychromatic light) was tested for its efficacy to treat SAD. In chronobiological terms this light is hypothesized to be more potent in inducing non-visual effects. In the present study fluorescent tubes that emit a high portion of short wavelength light on top of the normal wavelengths are tested for its superiority in treating SAD. This blue-enriched light (colour temperature 17000 ºK) is compared to standard light treatment (5000 º K) in SAD patients., The investigators hypothesise that blue- enriched light improve the therapeutic effects of light treatment leading to a higher response or the same response in a shorter time schedule compared to standard light treatment.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65;
* diagnosis of Seasonal affective Disorder, winter type according to DSM-IV;
* SIGH SAD rating higher then or equal to 18 on day 1;
* no other treatments for mood disorder during the study
* stay in the Netherlands during the study

Exclusion Criteria:

* other Axis 1 disorder according to DSM-IV
* acute suicide risk
* use of psychotropic drugs or photosensitizing drugs
* eye diseases other then usual effect of aging
* diabetes or epilepsy
* regular shift work

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2005-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
SIGH SAD depression observer rating | days 1, 8, 15, 22

SECONDARY OUTCOMES:
selfrating of depressive mood | once daily during 22 days

CONTACTS AND LOCATIONS:
Overall Officials: Y. Meesters, PhD, Study Chair — Department of Psychiatry, University Medical Center Groningen, The Netherlands
Locations (1):
- Department of Psychiatry, University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Gordijn MCM, 't Mannetje D, Meesters Y. The effects of blue-enriched light treatment compared to standard light treatment in Seasonal Affective Disorder. J Affect Disord. 2012 Jan;136(1-2):72-80. doi: 10.1016/j.jad.2011.08.016. Epub 2011 Sep 10. PMID 21911257